CLINICAL TRIAL: NCT00603044
Title: Mechanism of Action of Fluticasone Furoate in Childhood Obstructive Sleep Apnea Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15868B; 15868B
Record Dates: First submitted 2008-01-03; First posted 2008-01-28 (Estimated); Results first posted 2015-05-04 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Childhood Obstructive Sleep Apnea Syndrome (OSAS)
MeSH Terms: interventions — fluticasone furoate; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone furoate (Active Comparator): 55 mcg/nostril once daily for 2 weeks prior to adenotonsillectomy
  Interventions: Drug: fluticasone furoate
- No treatment (No Intervention)

INTERVENTIONS:
Drug: fluticasone furoate — treatment with fluticasone furoate (55 mcg/nostril once daily) for 2 weeks prior to adenotonsillectomy
  Other Names: Veramyst
  Arms: Fluticasone furoate

SUMMARY:
The purpose of this research is to find out how a nasal spray (fluticasone furoate), sometimes given to children with obstructive sleep apnea syndrome (OSAS), works on certain cells within a child's adenoids. We hypothesize that intranasal steroids lead to an upregulation of T regulatory cells in the adenoid tissues of children with OSAS. This will result in a local reduction in inflammation and edema explaining the improvement in OSAS.

DETAILED DESCRIPTION:
The objective was to determine the effect of intranasal corticosteroid therapy on T-regulatory cells and other inflammatory cytokines in adenoid tissues in children with obstructive sleep apnea syndrome.Children were randomized to either no treatment or treatment with fluticasone furoate nasal spray, 55 μg/nostril daily, for 2 weeks before adenotonsillectomy. Adenoid tissue was obtained at the time of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 2 and 12 years
* Polysomnogram results showing AHI >5/hr irrespective of saturations
* No other significant medical problems except well controlled asthma
* No chronic medication intake except bronchodilators and leukotriene receptor antagonists
* No systemic steroids within the past month
* No intranasal steroids within the past 2 weeks

Exclusion Criteria:

* Patients with OSAS who are overweight (BMI>95th percentile for age) or who have neurological or craniofacial abnormalities as these tend to have OSAS related to these factors per se.
* Females of the specified age group who have already had their first period.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fuad M Baroody, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- No Treatment: Subjects in this arm received no treatment.
Period: Overall Study
Arm/Group | Fluticasone Furoate | No Treatment
Started | 11 | 13
Completed | 11 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluticasone Furoate | No Treatment | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.24 (3.12) | 5.93 (3.32) | 5.62 (1.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of CD25 Pos/FoxP3 Positive Cells
Description: The number of tissue T-regulatory cells, as determined by staining with FOXP3, CD4, and CD25
Time Frame: following adenoidectomy (2 weeks)
Population: Some subjects were excluded due to technical issues.
Measure: Median (Full Range); unit: cells per High power field (HPF)
Arm/Group | Fluticasone Furoate | No Treatment
Number analyzed (Participants) | 11 | 10
cells per High power field (HPF) | 12.7 [3.1 to 35.2] | 14.6 [3.1 to 36.7]

2. Primary Outcome: Number of CD4 Pos/FOXP3 Positive Cells
Description: The number of tissue T-regulatory cells, as determined by staining with FOXP3, CD4, and CD25
Time Frame: following adenoidectomy (2 weeks)
Population: Some subjects were excluded due to technical issues.
Measure: Median (Full Range); unit: cells per High power field (HPF)
Arm/Group | Fluticasone Furoate | No Treatment
Number analyzed (Participants) | 11 | 10
cells per High power field (HPF) | 22.5 [3.3 to 38.8] | 21.4 [3.7 to 29.4]

3. Primary Outcome: IL-10 Staining Intensity
Description: IL-10 staining intensity on immunohistochemical staining of adenoid tissues. Units are Integrated optical density (IOD)/100 micrometer squared.
Time Frame: following adenoidectomy (2 weeks)
Population: Some subjects were excluded due to technical issues.
Measure: Mean (Standard Error); unit: IOD/100 micrometer squared
Arm/Group | Fluticasone Furoate | No Treatment
Number analyzed (Participants) | 9 | 10
IOD/100 micrometer squared | 437.4 (85.6) | 479.8 (6.0)

4. Primary Outcome: Amount of IL-10 Secreted by Adenoid Cells After PHA Stimulation
Description: Amount of IL-10 secreted by adenoid cells after PHA stimulation
Time Frame: following adenoidectomy (2 weeks)
Population: Some subjects were excluded due to technical issues.
Measure: Median (Full Range); unit: picogram per milliliter (pg/mL)
Arm/Group | Fluticasone Furoate | No Treatment
Number analyzed (Participants) | 11 | 12
picogram per milliliter (pg/mL) | 115 [6 to 204] | 210 [15 to 510]

5. Primary Outcome: Amount of TGF Secreted by Adenoid Cells After PHA Stimulation
Description: Amount of TGF secreted by adenoid cells after PHA stimulation
Time Frame: following adenoidectomy (2 weeks)
Population: Some subjects were excluded due to technical issues.
Measure: Median (Full Range); unit: picogram per milliliter (pg/mL)
Arm/Group | Fluticasone Furoate | No Treatment
Number analyzed (Participants) | 11 | 11
picogram per milliliter (pg/mL) | 944 [519 to 2555] | 906 [598 to 1071]

6. Secondary Outcome: Adjusted Volume of the Removed Adenoids
Description: To adjust for different weights of the children, the volume of the adenoids, estimated by water displacement in the operating room in mL, was divided by the respective weights (kg) of the patients and multiplied by 100.
Time Frame: following adenoidectomy (2 weeks)
Population: Some subjects were excluded due to technical issues.
Measure: Mean (Standard Error); unit: mL/kg x100
Arm/Group | Fluticasone Furoate | No Treatment
Number analyzed (Participants) | 10 | 9
mL/kg x100 | 13.0 (2.7) | 16.8 (3.8)

ADVERSE EVENTS:
Arm/Group | Fluticasone Furoate | No Treatment
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/13
Other Adverse Events (participants affected / at risk) | 0/11 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes